CLINICAL TRIAL: NCT00513344
Title: Efficacy of Polyphenols From Milk and Dark Chocolate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 06.38.MET
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-07

CONDITIONS: No Disease
Keywords: Endothelial function; Arterial stiffness; Dark chocolate; Milk chocolate; Polyphenols
MeSH Terms: interventions — Chocolate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- dark chocolate containing polyphenols (Experimental): dark chocolate
  Interventions: Dietary Supplement: Dark Chocolate
- Milk chocolate containing polyphenols (Experimental): Bespoke milk chocolate
  Interventions: Dietary Supplement: Milk Chocolate
- Control chocolate with no polyphenols (Active Comparator): cocoa-free chocolate
  Interventions: Dietary Supplement: Control (polyphenol-free) "Chocolate"

INTERVENTIONS:
Dietary Supplement: Dark Chocolate — 1 portion
  Arms: dark chocolate containing polyphenols
Dietary Supplement: Milk Chocolate — 1 portion
  Arms: Milk chocolate containing polyphenols
Dietary Supplement: Control (polyphenol-free) "Chocolate" — one portion
  Arms: Control chocolate with no polyphenols

SUMMARY:
Dark chocolate is one of the richest sources of polyphenols though it has been hypothesised that the bioavailability and therefore probably the bioefficacy of epicatechin from milk chocolate was reduced compared to dark. This study is designed to compare milk and dark chocolate as a source of polyphenols with a control "chocolate" for improving a risk biomarker for vascular disease.

DETAILED DESCRIPTION:
Dark chocolate is one of the richest sources of polyphenols, for example, a standard 40g portion of dark chocolate contains 400-800 mg of polyphenols, compared to red wine (170 mg /100ml) or an apple (200 mg/piece). Cocoa polyphenols, most notably the catechins, can exist in both lipid and water-based environments (amphipathic), meaning they can spare both lipophilic and hydrophilic vitamins. There have been a number of human trials conducted using chocolate or cocoa and measuring various endpoints. Most have been conducted with dark chocolate. An article in Nature found that the bioavailability of epicatechin from milk chocolate was substantially reduced compared to dark, and even dark taken with a glass of milk (Serafini et al 2003). The hypothesis was that the milk proteins bind to polyphenols, making them unavailable. Subsequent studies have not been able to reproduce this, but none have been conducted using solid chocolate as the first study, all have been done using a drink matrix, which may completely alter the binding interactions of the polyphenols and protein. To this end, this study is designed to compare solid chocolates as a source of polyphenols for improving a risk biomarker for vascular disease.

This study is designed as a blinded, three arm crossover trial. The primary outcome measure is to compare endothelial function after consumption of 3 chocolates (1 milk, 1 dark, 1 polyphenol-free control) with a secondary outcome of arterial stiffness. All volunteers will take all chocolate types in a crossover design. Subjects will undergo medical screening, anthropometry, physical activity and dietary assessments before randomization for the order of consumption.

ELIGIBILITY:
Inclusion Criteria:

* 25- 45 years, male and female
* Healthy as determined by the medical questionnaire
* Normal weight: BMI 19 - 25
* Having given informed consent

Exclusion Criteria:

* Intestinal or metabolic diseases/disorders such as diabetic, renal, hepatic, hypertension, pancreatic or ulcer, including lacto-intolerance.
* Have had a major gastrointestinal surgery.
* Have a regular consumption of medication.
* Have an exceptionally high intake of chocolate or similarly high polyphenol foods.
* Have a high and regular intake of vitamin supplements
* Have an alcohol intake: > 2 units a day
* Patient who cannot be expected to comply with treatment.
* Smoker
* Having a nut allergy
* Unwilling to consume chocolate
* Currently participating or having participated in another clinical trial during the last 3 weeks.
* Having given blood in the past three weeks
* More than 3 x 45 min of exercise per week

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Cooper, PhD, Principal Investigator — Société des Produits Nestlé (SPN); Gary Williamson, PhD, Study Director — Société des Produits Nestlé (SPN)
Locations (1):
- Nestle Research Center, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Heiss C, Finis D, Kleinbongard P, Hoffmann A, Rassaf T, Kelm M, Sies H. Sustained increase in flow-mediated dilation after daily intake of high-flavanol cocoa drink over 1 week. J Cardiovasc Pharmacol. 2007 Feb;49(2):74-80. doi: 10.1097/FJC.0b013e31802d0001. PMID 17312446
- [Background] Fisher ND, Hollenberg NK. Aging and vascular responses to flavanol-rich cocoa. J Hypertens. 2006 Aug;24(8):1575-80. doi: 10.1097/01.hjh.0000239293.40507.2a. PMID 16877960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 healthy subjects, 2 females and 3 males, were recruited within the staff of the Nestlé Research Center in June-July 2008.
Pre-assignment Details: From 3 days before the first test session no foods containing epicatechin or catechin or procyanidins should be ingested. The subjects received a single dose of the 3 products in a randomised order with a minimum of 3 days washout in between (crossover design). The duration of the study was a minimum of 15 days.
Groups:
- Each Subject Tested the Three Products Randomly Following: Before the 1st intervention, no food with polyphenols was admitted
  Each subject was administered the three products randomly(one product per one-day intervention) according to the six possible sequencies:
  * Either dark chocolate first, then milk chocolate then control
  * or dark chocolate first, then control, then milk chocolate
  * or control first, then dark chocolate, then milk chocolate
  * or Control first, then milk chocolate, then dark chocolate
  * or Milk chocolate first, then control, then dark chocolate
  * or milk chocolate first, then dark chocolate, then control r dark chocolate was given once in the morning (1 day) Products were administered in the morning of the testing day. The testing days (interventions) were separated by a three-day wash-out period.
Period: Diet Restriction (3 Days)
Arm/Group | Each Subject Tested the Three Products Randomly Following
Started | 5
Completed | 5
Not Completed | 0
Period: 1st Intervention 1 Day
Arm/Group | Each Subject Tested the Three Products Randomly Following
Started | 5
Completed | 5
Not Completed | 0
Period: Washout Period 3 Days
Arm/Group | Each Subject Tested the Three Products Randomly Following
Started | 5
Completed | 5
Not Completed | 0
Period: 2nd Intervention 1 Day
Arm/Group | Each Subject Tested the Three Products Randomly Following
Started | 5
Completed | 5
Not Completed | 0
Period: Washout Period 3 Days
Arm/Group | Each Subject Tested the Three Products Randomly Following
Started | 5
Completed | 5
Not Completed | 0
Period: 3rd Intervention 1 Day
Arm/Group | Each Subject Tested the Three Products Randomly Following
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive control first, milk chocolate first, and dark chocolate first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 34 (7)
Age, Customized [Number; unit: participants]
  <= 28 years | 0
  between 28 and 42 years | 5
  >= 42 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  Switzerland | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Reactive Hyperemia Index (RHI) From Baseline (20 Min Before Product Intake) to 2 Hours Following Product Intake
Description: Value of RHI at 2 hours minus value at baseline. RHI reflects the endothelial function of a vessel at the distal phalanx of a finger, i.e. the capacity of the vessel to dilate after an ischemia. RHI is the increase of blood flow following the occlusion of the brachial artery during 5 minutes by the inflation of an armcuff. RHI was measured by peripheral arterial tonometry using a fingerprobe connected to an EndoPat analyser.
Time Frame: Baseline and 2 hours
Population: Taking into account the fact that there is no background data and that we need to have accurate evaluation of central tendency and dispersion, a minimum of five complete subjects are needed.
  Data from all randomized subjects were considered in the intention to treat model (for the primary outcome).
Measure: Mean (Standard Error); unit: percentage of the pulse wave amplitude
Groups:
- Control Chocolate With no Polyphenols: cocoa-free chocolate
  Control (polyphenol-free)
- Milk Chocolate Containing Polyphenols: Bespoke milk chocolate
  Milk Chocolate : 1 portion
- Dark Chocolate Containing Polyphenols: dark chocolate
  Dark Chocolate : 1 portion
Arm/Group | Control Chocolate With no Polyphenols | Milk Chocolate Containing Polyphenols | Dark Chocolate Containing Polyphenols
Number analyzed (Participants) | 5 | 5 | 5
percentage of the pulse wave amplitude | 2.12 (0.52) | 2.30 (0.71) | 2.26 (0.65)

2. Secondary Outcome: Change in Arterial Stiffness From Baseline (20 Min Before Product Intake) to Two Hours Following Product Intake
Description: Value of arterial stiffness at 2 hours minus value at baseline. Arterial stiffness is also automatically calculated by peripheral arterial tonometry which consists in measuring the peripheral vessel endothelial response to an ischemia provoked by a 5-min occlusion of the humeral artery using an armcuff.
  An increase in arterial stiffness means an increase in the resistance of the vessel wall which reflects an impaired endothelial response to ischemia.
Time Frame: baseline and 2 hours
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Control Chocolate With no Polyphenols | Milk Chocolate Containing Polyphenols | Dark Chocolate Containing Polyphenols
Number analyzed (Participants) | 5 | 5 | 5
percentage of baseline | -13.23 (11.16) | 1.23 (12.87) | -9.49 (15.03)

ADVERSE EVENTS:
Description: Adverse Events Not Collected
Arm/Group | Dark Chocolate | Milk Chocolate | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes